CLINICAL TRIAL: NCT05132413
Title: A Phase 3, Randomized Double-blind, Placebo-controlled, Multicenter Study of SHR-1701 in Combination With Bevacizumab and Chemotherapy in Advanced or Metastatic Non-squamous Non-small-cell Lung Cancer With EGFR Mutation After Failure of TKIs
Brief Title: A Study of SHR-1701 Plus Bevacizumab and Chemotherapy in Non-Small-Cell-Lung-Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1701-III-310
Record Dates: First submitted 2021-11-12; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Advanced or Metastatic Non-squamous Non-small-cell Lung Cancer
MeSH Terms: interventions — SHR-1701; Pemetrexed; Cisplatin; Carboplatin; Bevacizumab

STUDY DESIGN:
Intervention Model Description: SHR-1701/ Placebo Plus Chemotherapy With or Without Bevacizumab
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- treatment group (Experimental)
  Interventions: Drug: SHR-1701 + Pemetrexed Disodium + cisplatin/carboplatin + bevacizumab
- Placebo group 1 (Placebo Comparator)
  Interventions: Drug: Placebo + SHR-1701 + Pemetrexed Disodium+ cisplatin/carboplatin
- Placebo group 2 (Placebo Comparator)
  Interventions: Drug: Placebo 1 + Placebo 2 +Pemetrexed Disodium + cisplatin/carboplatin

INTERVENTIONS:
Drug: SHR-1701 + Pemetrexed Disodium + cisplatin/carboplatin + bevacizumab — SHR-1701 + Pemetrexed Disodium + cisplatin/carboplatin + bevacizumab
  Arms: treatment group
Drug: Placebo + SHR-1701 + Pemetrexed Disodium+ cisplatin/carboplatin — Placebo + SHR-1701 + Pemetrexed Disodium+ cisplatin/carboplatin
  Arms: Placebo group 1
Drug: Placebo 1 + Placebo 2 +Pemetrexed Disodium + cisplatin/carboplatin — Placebo 1 + Placebo 2 +Pemetrexed Disodium + cisplatin/carboplatin
  Arms: Placebo group 2

SUMMARY:
Evaluate efficacy and safety of SHR-1701 in combination with bevacizumab and chemotherapy in advanced or metastatic non-squamous non-small-cell lung cancer with EGFR mutation after failure of TKIs

ELIGIBILITY:
Inclusion Criteria:

-

A subject must satisfy all of the following criteria to be considered for inclusion in the study:

1. Histologically or cytologically confirmed advanced or metastatic non-squamous non-small cell lung cancer.
2. Failed with prior EGFR-TKIs treatments.
3. Measurable disease, as defined by RECIST v1.1
4. The Eastern Cancer Cooperative Group (ECOG) performance status of 0 or 1
5. Life expectancy ≥ 3 months
6. Adequate hematologic and end-organ function as defined in the protocol

Exclusion Criteria:

-

A subject who meets any of the following criteria will be excluded from study entry:

1. Histologically or cytologically confirmed mixed SCLC and NSCLC.
2. Symptomatic, untreated or active central nervous system metastases.
3. Systemic therapy with immunosuppressive agents within 2 weeks prior to initiation of study treatment
4. With any active autoimmune disease or history of autoimmune disease.
5. Inadequately controlled hypertension.
6. Tumour infiltration into the great vessels on imaging.
7. History of haemoptysis ≥2.5ml per episode within 1 month prior to initiation of study treatment.
8. Uncontrolled tumour-related pain.
9. Patients with active hepatitis B or hepatitis C
10. Severe infections within 4 weeks prior to initiation of study treatment. Active tuberculosis within one year prior to initiation of study treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 561 (Estimated)
Dates: Start 2021-12-30 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs), serious adverse events (SAEs), and immune-related adverse events (irAEs) as per NCI-CTC AE 5.0 （Stage I） | 2 years
BIRC-assessed progression-free survival (PFS) as per RECIST v1.1（Stage II） | 2 years

SECONDARY OUTCOMES:
Progression free survival (PFS)（Stage I） | 2 years
Objective response rate (ORR)（Stage I） | 2 years
Disease control rate (DCR) （Stage I） | 2 years
Duration of response (DOR) （Stage I） | 2 years
Overall survival (OS) （Stage I） | 2 years
Progression free survival (PFS)（Stage II） | 2 years
Objective response rate (ORR)（Stage II） | 2 years
Disease control rate (DCR)（Stage II） | 2 years
Duration of response (DOR) （Stage II） | 2 years
Overall survival (OS) （Stage II） | 2 years
Incidence and severity of adverse events (AEs), serious adverse events （Stage II） | 2 years
(SAEs), and immune-related adverse events (irAEs) as per NCI-CTC AE 5.0（Stage II） | 2 years

IPD SHARING:
Plan to Share IPD: Undecided